CLINICAL TRIAL: NCT04809285
Title: Use of the Guardian™ Connect System With Smart Connected Devices
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Diabetes (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CIP331
Record Dates: First submitted 2021-03-18; First posted 2021-03-22 (Actual); Results first posted 2024-12-10 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-11

CONDITIONS: Type 1 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Guardian™ Connect system, InPen™ Basal smart cap, and smart insulin pens (Experimental): All subjects will wear the Guardian Connect system (real-time continuous glucose monitoring (CGM)) continuously and use smart insulin pens or insulin pens with smart caps for multiple daily injections and continue their standard therapy throughout the duration of the study.
  Interventions: Device: Guardian™ Connect system, InPen™ Basal smart cap, smart insulin pens, and InPen™ Diabetes Management app

INTERVENTIONS:
Device: Guardian™ Connect system, InPen™ Basal smart cap, smart insulin pens, and InPen™ Diabetes Management app — Guardian™ Connect system consists of Guardian™ Connect app, Guardian™ Connect transmitter, and Guardian Sensor (3), will be working with InPen™ Basal smart cap and smart insulin pens and InPen™ Diabetes Management app for multiple daily injections. The subject's insulin delivery, sleep, physical activity (as applicable), food intake data, and medication (as applicable) will be collected through applications with meal logging and medication requiring manual entry. In addition, subjects may also participate in optional self-administered insulin injection video capture and upload using a secure cloud-based site and/or monthly menstrual cycle logging using Apple Health and/or cardiac monitoring using BodyGuardian MINI.

SUMMARY:
The purpose of this study is to collect sensor, insulin, sleep, activity and food/meal data for a minimum of 90 days of device wear (Phase 1) and up to a maximum of 9 months of device wear (Phase 2) with optional insulin injection video capture and/or menstrual cycle tracking and/or cardiac monitoring in subjects with insulin requiring diabetes 2-80 years of age.

DETAILED DESCRIPTION:
The study is a multi-center, prospective single-arm design without controls. All subjects will participate for a minimum of 90 days (Phase 1) and some subjects 18 years of age or older will participate for up to 9 months (Phase 2). All subjects will wear the Guardian Connect system (real-time continuous glucose monitoring (CGM)) continuously and use smart insulin pens or insulin pens with smart caps for multiple daily injections and continue their standard therapy throughout the duration of the study.

The subject's insulin delivery, sleep, physical activity (as applicable), food intake data, and medication (as applicable) will be collected through applications with meal logging and medication requiring manual entry. In addition, subjects may also participate in optional self-administered insulin injection video capture and upload using a secure cloud-based site and/or monthly menstrual cycle logging using Apple Health and/or cardiac monitoring using BodyGuardian MINI.

ELIGIBILITY:
Inclusion Criteria

1. Individual is 2-80 years of age at time of consent.
2. A clinical diagnosis of type 1 or type 2 diabetes as determined by investigator for:

   * at least the last 6 months for subjects 2-6 years of age
   * at least the last 12 months for subjects 7-80 years of age
3. Subject is on multiple daily injection therapy (3 or more insulin injections per day one of which is a long acting insulin injection), is currently using or is willing and can afford to use insulin pen(s) and pen cartridge(s).
4. Subject is currently using or is willing to use the Guardian Connect system during the study.
5. Subject agrees to comply with the study protocol requirements.
6. For adult subjects: Subject is capable of providing legal consent without a legal authorized representative.

Exclusion Criteria

1. Subject is using a syringe and unwilling or unable to use insulin pen(s).
2. Subject is using an insulin pump.
3. Subject is currently using a non-Medtronic standalone CGM system and unwilling to use only the Guardian Connect system during the study.
4. Subject is using hydroxyurea at time of screening or plans to use it during the study.
5. Subject will not tolerate tape adhesive in the area of device placement as assessed by a qualified provider.
6. Subject has any unresolved adverse skin condition in the area of device placement (e.g. psoriasis, rash, Staphylococcus infection).
7. Subject is actively participating in or plans to enroll in an investigational study (e.g. drug or device), other than this study, wherein they have received treatment from an investigational drug or device.
8. Subject has a positive urine pregnancy test at time of screening.
9. Subject is female, sexually active without the use of contraception, able to become pregnant or plans to become pregnant during the course of the study.
10. Subject is unwilling to participate in study procedures.
11. Subject is directly involved in the study as research staff.

Ages: 2 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 217 (Actual)
Dates: Start 2021-04-06 (Actual); Primary Completion 2023-09-29 (Actual); Study Completion 2023-09-29 (Actual)

CONTACTS AND LOCATIONS:
Locations (14):
- United States (14):
  - Arkansas Diabetes and Endocrinology Center, Little Rock, Arkansas
  - Loma Linda University Medical Center, Loma Linda, California
  - Mary and Dick Allen Diabetes Center, Newport Beach, California
  - Salinas Valley Memorial Healthcare System, Salinas, California
  - Barbara Davis Center for Childhood Diabetes, Aurora, Colorado
  - Atlanta Diabetes Associates, Atlanta, Georgia
  - Endocrine Research Solutions, Inc., Roswell, Georgia
  - Rocky Mountain Diabetes and Osteoporosis Center, Idaho Falls, Idaho
  - Endocrine and Metabolic Consultants, Rockville, Maryland
  - Rhode Island Hospital (Lifespan Clinical Research Center), Providence, Rhode Island
  - AM Diabetes and Endocrinology Center, Bartlett, Tennessee
  - Texas Diabetes and Endocrinology, Austin, Texas
  - Texas Diabetes and Endocrinology, Round Rock, Texas
  - Rainer Clinical Research Center, Renton, Washington

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All subjects participated for a minimum of 90 days (Phase 1) and some subjects 18 years of age or older participated for up to 9 months (Phase 2). All subjects wore the Guardian Connect system (real-time CGM) continuously and used smart insulin pens or insulin pens with smart caps for multiple daily injections and continued their standard therapy throughout the duration of the study.
Period: Phase 1
Arm/Group | Guardian™ Connect System, InPen™ Basal Smart Cap, and Smart Insulin Pens
Started (Excludes 9 subjects who were screen failures) | 208
Completed | 168
Not Completed | 40
Not completed — Lost to Follow-up | 6
Not completed — Protocol Violation | 2
Not completed — Physician Decision | 3
Not completed — Withdrawal by Subject | 29
Period: Phase 2
Arm/Group | Guardian™ Connect System, InPen™ Basal Smart Cap, and Smart Insulin Pens
Started | 67 (Not all subjects that completed Phase 1 opted to/were eligible to participate in Phase 2)
Completed | 60
Not Completed | 7
Not completed — Protocol Violation | 3
Not completed — Withdrawal by Subject | 4

BASELINE CHARACTERISTICS:
Population: Number of subjects who enrolled into study at Phase 1
Arm/Group | Guardian™ Connect System, InPen™ Basal Smart Cap, and Smart Insulin Pens
Number analyzed (Participants) | 208
Age, Continuous [Mean (Standard Deviation); unit: Years] — Population: One subject (out of the 208 enrolled) did not provide this information during their study visit.
  Years
    number analyzed (Participants) | 207
    (all) | 37.3 (17.8)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: One subject (out of the 208 enrolled) did not provide this information during their study visit.
  Participants
    number analyzed (Participants) | 207
    Female | 97
    Male | 110
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: One subject (out of the 208 enrolled) did not provide this information during their study visit.
  Participants
    number analyzed (Participants) | 207
    Hispanic or Latino | 38
    Not Hispanic or Latino | 168
    Unknown or Not Reported | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: One subject (out of the 208 enrolled) did not provide this information during their study visit.
  Participants
    Race: number analyzed (Participants) | 207
    Race: White | 154
    Race: Asian | 13
    Race: American Indian or Alaska Native | 1
    Race: American Indian or Alaska Native, Black or African American, White | 2
    Race: American Indian or Alaska Native, White | 1
    Race: Black or African American | 28
    Race: Other | 8
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 208

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Time in Hypoglycemia
Description: The overall mean percentage of time in hypoglycemia (SG < 70 mg/dL)
Time Frame: Day 1 to Day 90 in Phase 1 and Day 91 to up to 9 months in Phase 2
Population: The number of participants analyzed reflects the number of subjects for which any data were available.
Measure: Mean (Standard Deviation); unit: percentage of time
Groups:
- Phase 1: Subjects who participated in Phase 1 of the study.
- Phase 2: Subjects who participated in Phase 2 of the study (some subjects 18 years of age or older who participated for up to 9 months after participating in Phase 1).
Arm/Group | Phase 1 | Phase 2
Number analyzed (Participants) | 192 | 63
percentage of time | 3.1 (3.4) | 2.7 (3.3)

2. Primary Outcome: Percentage of Time in Euglycemia
Description: The overall mean percentage of time in euglycemia (SG 70-180 mg/dL)
Time Frame: Day 1 to Day 90 in Phase 1 and Day 91 to up to 9 months in Phase 2
Population: The number of participants analyzed reflects the number of subjects for which any data were available.
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | Phase 1 | Phase 2
Number analyzed (Participants) | 192 | 63
percentage of time | 59.5 (20.2) | 58.7 (20.0)

3. Primary Outcome: Percentage of Time in Hyperglycemia
Description: The overall mean percentage of time in hyperglycemia (SG > 180 mg/dL)
Time Frame: Day 1 to Day 90 in Phase 1 and Day 91 to up to 9 months in Phase 2
Population: The number of participants analyzed reflects the number of subjects for which any data were available.
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | Phase 1 | Phase 2
Number analyzed (Participants) | 192 | 63
percentage of time | 37.5 (20.9) | 38.7 (20.7)

ADVERSE EVENTS:
Time Frame: Day 1 to Day 90 in Phase 1 and Day 91 to up to 9 months in Phase 2
Arm/Group | Phase 1 | Phase 2
All-Cause Mortality (participants affected / at risk) | 0/208 | 0/67
Serious Adverse Events (participants affected / at risk) | 5/208 | 3/67
Other Adverse Events (participants affected / at risk) | 20/208 | 0/67
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1 (N=208) | Phase 2 (N=67)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Angina unstable (Cardiac disorders) | 0 (0) | 1 (1)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Hypothermia (General disorders) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Substance abuse (Psychiatric disorders) | 1 (1) | 0 (0)
End stage renal disease (Renal and urinary disorders) | 1 (1) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1 (N=208) | Phase 2 (N=67)
Medical device pain (General disorders) | 1 (1) | 0 (0)
Medical device site dermatitis (General disorders) | 4 (4) | 0 (0)
Medical device site discolouration (General disorders) | 2 (2) | 0 (0)
Medical device site haemorrhage (General disorders) | 1 (1) | 0 (0)
Medical device site irritation (General disorders) | 7 (7) | 0 (0)
Medical device site pruritus (General disorders) | 4 (4) | 0 (0)
Medical device site rash (General disorders) | 3 (3) | 0 (0)
Medical device site vesicles (General disorders) | 1 (1) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0)
Skin abrasion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2021-06-08): https://cdn.clinicaltrials.gov/large-docs/85/NCT04809285/Prot_000.pdf
  • Statistical Analysis Plan (2022-01-13): https://cdn.clinicaltrials.gov/large-docs/85/NCT04809285/SAP_001.pdf